CLINICAL TRIAL: NCT04168489
Title: Based on Functional Magnetic Resonance Imaging Technology to Evaluate the Analgesic Effect of TMS on Primary Dysmenorrhea and Neuroimaging Prediction Study
Brief Title: Evaluation of the Effect of TMS on Primary Dysmenorrhea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Grant Nos. 81901723
Record Dates: First submitted 2019-10-25; First posted 2019-11-19 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Primary Dysmenorrhea
Keywords: rTMS; Primary Dysmenorrhea

STUDY DESIGN:
Intervention Model Description: (a) consistent with the diagnostic criteria for primary dysmenorrhea according to the American College of Obstetricians and Gynecologists; (b) regular menstrual cycles (27-32 days); and (c) the average intensity of dysmenorrhoeic pain in the past 6 months should be rated ≥4 on a visual analogue scale (VAS) (0 = no pain, 10 = the worst imaginable pain).
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active rTMS (Active Comparator)
  Interventions: Device: active rTMS
- sham rTMS (Sham Comparator)
  Interventions: Device: sham rTMS

INTERVENTIONS:
Device: active rTMS — (rTMS) is received preliminary approval because of its noninvasive and safe analgesic effect.
  Arms: active rTMS
Device: sham rTMS — The sham rTMS is inactive and similar to placebo effect.
  Arms: sham rTMS

SUMMARY:
Based on the pain threshold and visual simulation score, primary dysmenorrhea patients will be divided into treatment effective group or non-effective group.According to the functional magnetic resonance imaging, the investigators investigate whether there is characteristic or secondary brain features before and after rTMS intervention.

DETAILED DESCRIPTION:
Long term primary dysmenorrhea may induce a series of disorders involving psychology, lower quality of life, or even developing chronic organic lesion or chronic pain. Effective symptom improvement is urgently needed. During the Non-pharmaceutical interventions, repetitive transcranial magnetic stimulation (rTMS) is received preliminary approval because of its noninvasive and safe analgesic effect. In this randomized single blind longitudinal study, the investigators investigate the analgesic effect of rTMS in long term moderate-to-severe primary dysmenorrhea women. Based on the pain threshold and visual simulation score, primary dysmenorrhea patients will be divided into treatment effective group or non-effective group. According to the functional magnetic resonance imaging, the investigators investigate whether there is characteristic or secondary brain features before and after rTMS intervention. By combining pre and post performances of the degree of dysmenorrhea, behavioral data and sensitive hematological indicators, the investigators intend to build an association model between brain and pain development curve. Using correlation and multiple regression analysis method, the investigators intend to find sensitive neuroimaging biomarkers in predicting the analgesic effect of rTMS. The current study is not only contributing to improve the central nervous systematic mechanism of rTMS in chronic pelvic pain, but also significant for clinical effective treatment based on neuroimaging predictive markers.

ELIGIBILITY:
Inclusion Criteria:

* consistent with the diagnostic criteria for primary dysmenorrhea according to the American College of Obstetricians and Gynecologists;
* regular menstrual cycles (27-32 days);
* the average intensity of dysmenorrhoeic pain in the past 6 months should be rated ≥4 on a visual analogue scale (VAS) (0 = no pain, 10 = the worst imaginable pain).

Exclusion Criteria:

* organic pelvic disease;
* using oral contraceptives, hormonal supplements, Chinese traditional medicine or any central-acting medication (e.g., opioids, anti-epileptics) within 6 months before the study;
* comorbid chronic pain states;
* alcohol, nicotine or drug addiction;
* neurologic disease or psychiatric disorder;
* history of childbirth;
* a positive pregnancy test or immediate plans for pregnancy;
* any MRI contraindications. In addition, no analgesics were consumed 24 hours prior to the experiment.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of effect of rTMS for primary dysmenorrhea | From 1 month before treatment to 3 months after treatment for each volunteers(through study completion, an average of 2 years)
  Assessments using Visual Analog Score for pain(Units on a Scale) in primary dysmenorrhea during menstrual phase to evaluate the effect of rTMS

CONTACTS AND LOCATIONS:
Overall Officials: wanghuan Dun, M.D., Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi, China